CLINICAL TRIAL: NCT02596204
Title: Diabetes Care Transformation: Diabetes Data Registry and Intensive Remote Monitoring
Acronym: DCT1A
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospitals and Clinics of Minnesota (Other)
Collaborators: UnitedHealth Group (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1506-073
Record Dates: First submitted 2015-10-05; First posted 2015-11-04 (Estimated); Last update posted 2017-08-01 (Actual); Status verified 2017-07

CONDITIONS: Type 1 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Data Upload (Active Comparator): Subjects will wear a FitBit activity monitor and continue to use their insulin pump. FitBit, pump and sensor (if applicable) data will be uploaded at least weekly. Subjects will continue to receive usual diabetes care. Phone calls and emails to the diabetes clinic will be initiated by the family.
  Interventions: Device: FitBit
- Weekly Review (Experimental): Subjects will wear a FitBit activity monitor and continue to use their insulin pump. FitBit, pump and sensor (if applicable) data will be uploaded at least weekly. For subjects in the weekly review group, research staff (diabetes educator, nurse practitioner and/or physician) will review uploaded blood glucose, pump, and available sensor, activity and sleep data on a weekly basis. If glucose patterns are identified which suggest a change to diabetes management (ie insulin dose changes), the family will be contacted by text, email or telephone to review glucose patterns and to review staff recommendations.
  Interventions: Other: Weekly Review; Device: FitBit

INTERVENTIONS:
Other: Weekly Review — Subjects will wear a FitBit activity monitor and continue to use their insulin pump. Fitbit, pump and sensor (if applicable) data will be uploaded at least weekly. For subjects in the weekly review group, research staff (CDE, NP and/or MD) will review uploaded blood glucose, pump, and available sensor, activity and sleep data on a weekly basis. If glucose patterns are identified which suggest a change to diabetes management (ie insulin dose changes), the family will be contacted by text, email or telephone to review glucose patterns and to review staff recommendations.
  Arms: Weekly Review
Device: FitBit — All subjects will wear a FitBit activity monitor.

SUMMARY:
With emerging mobile technology, sharing glucose, insulin and sensor data with the clinic for frequent and timely monitoring is now feasible. The investigators propose to leverage this new technology to provide children and families with appropriate interventions to help manage their diabetes.

DETAILED DESCRIPTION:
The investigators will collect insulin dosing via pump records, blood glucose meter, continuous glucose sensor, activity, heart rate, and sleep data on a weekly basis from 100 children with diabetes. The investigators hypothesize that with the collection and analysis of insulin, blood glucose, sensor, activity, heart rate and sleep data in children with diabetes the investigators can identify glucose patterns and predictors of acute events.

The 100 children will be randomized to either conventional therapy (data upload group) or intensive remote therapy (weekly review group). Conventional therapy will consist of routine quarterly visits to the clinic and as-needed communication with the diabetes staff, initiated by the family, between study visits. Intensive remote therapy will consist of routine quarterly visits to the clinic along with weekly remote review of insulin and blood glucose data by the research staff, and additional communication with the family, initiated by the diabetes staff as needed, between visits. The investigators hypothesize that with weekly, manual review of real-time insulin, glucose, and activity data in children with diabetes, and recommended regimen changes based on the data, the investigators will be able to lower HbA1c values in children in the weekly review group as compared to children in the data upload group.

ELIGIBILITY:
Inclusion Criteria:

1. Type 1 diabetes, using an insulin pump (Medtronic, Omnipod, Animas)
2. Duration of diabetes >1 year
3. Age: 8-17 years of age, inclusive.
4. Hemoglobin A1c 8.0-10.0% at baseline visit, inclusive.
5. Seen in the McNeely Diabetes Clinic within the past 6 months.
6. The family/child is testing blood glucose at least 4 times a day.
7. The family has a smart phone and service.

Exclusion Criteria:

1. The child is not using insulin for management of diabetes.
2. The child uses multiple daily injections of insulin.
3. The child is unwilling to use the wearable device, or the family is unwilling or unable to upload glucose and insulin data on a routine basis
4. The family is unwilling or unable to upload data from devices such as meter, pump, sensor, wearable device.
5. Diagnosis of a mental health disorder.
6. Parent/child does not speak English as the device software is only available in English.

Ages: 8 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 113 (Actual)
Dates: Start 2015-09; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Change in Hemoglobin A1c | From baseline to 6 months
  Change in HbA1c from baseline to 6 months

SECONDARY OUTCOMES:
Health care utilization | 6 months
  The investigators will track the number of phone calls to clinic, emergency department visits and hospitalizations over 6 months between data upload and weekly review groups
PedsQL Inventory (PedsQL) | 6 months
  The investigators will assess change in the PedsQL (Peds Quality of Life) Inventory from baseline to 6 months between data upload and weekly review groups.
Diabetes Family Conflict Scale (DFCS) | 6 months
  The investigators will assess change in the Diabetes Family Conflict Scale from baseline to 6 months between data upload and weekly review groups.
Center for Epidemiology Scale- Depression (CES-D) survey | 6 months
  The investigators will assess change in the Center for Epidemiology Scale- Depression from baseline to 6 months between data upload and weekly review groups.
Problem Areas in Diabetes (PAID) survey | 6 months
  The investigators will assess change in the Problem Areas in Diabetes- pediatrics and Problem Areas in Diabetes- parent from baseline to 6 months between data upload and weekly review groups.
Change in Hemoglobin A1c | Change from 6 months to 9 months
  Change in hemoglobin A1c from 6 months (end of active intervention) to 9 months

CONTACTS AND LOCATIONS:
Locations (1):
- Children's Hospitals and Clinics of Minnesota, Saint Paul, Minnesota, United States